CLINICAL TRIAL: NCT04498741
Title: A Non-Randomized, Open-Label, Three-Part, Drug-Drug Interaction Study to Evaluate the Effects of EDP-938 on the Pharmacokinetics of Tacrolimus, Dabigatran, Rosuvastatin and Midazolam in Healthy Subjects
Brief Title: Drug-Drug Interaction Study Between EDP-938, Tacrolimus, Dabigatran, Rosuvastatin and Midazolam in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Collaborators: Pharmaceutical Research Associates (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EDP 938-006
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2020-08

CONDITIONS: RSV Infection
Keywords: drug-drug interaction
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — EDP-938; Tacrolimus; Dabigatran; Rosuvastatin Calcium; Midazolam

STUDY DESIGN:
Intervention Model Description: 4-Part Single Group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- EDP-938 and tacrolimus interaction (Part 1) (Experimental)
  Interventions: Drug: EDP-938; Drug: Tacrolimus
- EDP-938 and dabigatran interaction (Part 2) (Experimental)
  Interventions: Drug: EDP-938; Drug: Dabigatran
- EDP-938 and rosuvastatin interaction (Part 3) (Experimental)
  Interventions: Drug: EDP-938; Drug: Rosuvastatin
- EDP-938 and midazolam interaction (Part 4) (Experimental)
  Interventions: Drug: EDP-938; Drug: Midazolam

INTERVENTIONS:
Drug: EDP-938 — Subjects will receive EDP-938 once daily on Days 10 through 27 (Part 1)
  Arms: EDP-938 and tacrolimus interaction (Part 1)
Drug: EDP-938 — Subjects will receive EDP-938 once daily on Days 5 through 15 (Part 2)
  Arms: EDP-938 and dabigatran interaction (Part 2)
Drug: EDP-938 — Subjects will receive EDP-938 once daily on Days 5 through 15 (Part 3)
  Arms: EDP-938 and rosuvastatin interaction (Part 3)
Drug: Tacrolimus — Subjects will receive tacrolimus once daily on Day 1 and Day 24
  Arms: EDP-938 and tacrolimus interaction (Part 1)
Drug: Dabigatran — Subjects will receive dabigatran once daily on Day 1 and Day 13
  Arms: EDP-938 and dabigatran interaction (Part 2)
Drug: Rosuvastatin — Subjects will receive rosuvastatin once daily on Day 1 and Day 13
  Arms: EDP-938 and rosuvastatin interaction (Part 3)
Drug: EDP-938 — Subjects will receive EDP-938 once daily on Days 3 through 16 (Part 4)
  Arms: EDP-938 and midazolam interaction (Part 4)
Drug: Midazolam — Subjects will receive midazolam once daily on Day 1 and Day 16
  Arms: EDP-938 and midazolam interaction (Part 4)

SUMMARY:
A Non-Randomized, Open-Label, Three-Part, Drug-Drug Interaction Study to Evaluate the Effects of tacrolimus, dabigatran, rosuvastatin and midazolam on the Pharmacokinetics and Safety of EDP-938 in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject.
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 55 years, inclusive.
* Screening body mass index (BMI) of 18 to 30 kg/m2 with a minimum body weight of 50 kg
* Female subjects of childbearing potential must agree to use two effective methods of contraception from the date of Screening until 90 days after the last dose of EDP 938.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease
* Pregnant or nursing females.
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.
* A positive urine drug screen at Screening or Day -1.
* Current tobacco smokers or use of tobacco within 3 months prior to Screening.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy).
* History of regular alcohol consumption.
* Participation in a clinical trial within 30 days prior to the first dose of study drug.
* For Part 1 subjects:
* Clinical history or evidence at Screening consistent with hyperkalemia, hypertension and/or diabetes mellitus
* For Part 2 Subjects:
* Clinical history or evidence at screening of medically significant bleeding
* History of a mechanical heart valve placement, a thromboembolic event or clinically significant thrombotic event, an autoimmune disease, eg, systemic lupus erythematosus (SLE), or recurrent spontaneous abortions
* A platelet count <LLN, or INR >ULN, or aPTT > ULN at Screening
* Ongoing daily use of nonsteroidal anti-inflammatory drugs
* For Part 3 subjects:
* AST and/or ALT >ULN at Screening
* For Part 4 subjects:
* History of glaucoma

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Cmax of tacrolimus with and without coadministration with EDP-938 | up to 29 days
AUC of tacrolimus with and without coadministration with EDP-938 | up to 29 days
Cmax of dabigatran with and without coadministration with EDP-938 | up to 17 days
AUC of dabigatran with and without coadministration with EDP-938 | up to 17 days
Cmax of rosuvastatin with and without coadministration with EDP-938 | up to 17 days
AUC of rosuvastatin with and without coadministration with EDP-938 | up to 17 days
Cmax of midazolam with and without coadministration with EDP-938 | up to 17 days
AUC of midazolam with and without coadministration with EDP-938 | up to 17 days

SECONDARY OUTCOMES:
Safety measured by adverse events | up to 34 days

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- Pharmaceutical Research Associates, Inc.,, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No